CLINICAL TRIAL: NCT01655914
Title: Open Label, Randomized, Three-way Crossover Study to Assess the Safety and the Pharmacokinetics of Sublingual Flumazenil (CRLS035) in Healthy Adults
Brief Title: Safety and Pharmacokinetic Study of Sublingual Flumazenil (CRLS035) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Coeruleus Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CRLS002
Record Dates: First submitted 2012-07-30; First posted 2012-08-02 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Flumazenil

ARMS (2):
- Arm A (Active Comparator): Sequence of Exposure:
  Sequence A (N=5) Week 1: S/L 1.1 mg Week 2: S/L 2.2 mg Week 3: IV 0.2 mg Week 4: S/L 2.2 mg with 240 ml water
  Interventions: Drug: Flumazenil
- Arm B (Active Comparator): Sequence B (N=5) Week 1: IV 0.2 mg Week 2: S/L 2.2 mg Week 3: S/L 1.1 mg Week 4: S/L 2.2 mg with high fat diet
  Interventions: Drug: Flumazenil

INTERVENTIONS:
Drug: Flumazenil

SUMMARY:
This study compare the pharmacokinetic (PK) profile of sublingual CRLS035 (two doses) to I.V flumazenil administration.

Selection of study drug dosage: CRLS035 - sublingual Flumazenil will be administrated at a final dosage of 1.1 mg per 100 µl and 2.2 mg (200 µl) in a sublingual spray administration.

Currently, Flumazenil is given as an IV drug with a repetitive administration of doses of 0.2 mg up to 3 mg per hour. As the bioavailability of Flumazenil is expected to be lower than the IV administration, 1.1 mg and 2.2 mg will be tested in sublingual delivery. The suggested doses in this study are very safe according to the following data: first, sublingual and buccal administration of Flumazenil have been detailed previously with similar and higher doses with no side effects, secondly, IV dose may reach 3 mg and thirdly, oral administration has been reported as up to 600 mg/dose.

The purpose of this study is to determine the single dose PK profile of SL CRLS035. This study is designed to collect short-term safety data and to monitor the PK profile of CRLS035.

Primary Objective The primary objective is to determine the single dose safety and PK profile of SL CRLS035 using the marketed IV flumazenil formulation as the comparator.

Secondary Objectives The secondary objectives are to (1) characterize the concentration time course of two dose levels of SL CRLS035 to support dose selection for Phase 2 and 3 studies and to evaluate the safety and tolerability of flumazenil formulations; (2)To evaluate the effect of high fat diet and water consumption on the PK profile.

ELIGIBILITY:
Inclusion Criteria:

1. The subject understood and voluntarily signed an informed consent form prior to any study-mandated procedure.
2. Male or female aged ≥18-at screening.
3. Body mass index ≥ 18.5 and < 32 kg/m2.
4. Subject is in good health as determined by a medical history, physical examination and ECG.
5. Negative any use of illicit drug, alcohol (ethanol), stimulants.

Exclusion Criteria:

1. Any use of medications within 1 month prior to screening visit, except for contraceptive pills.
2. Previous exposure to Benzodiazepines and/or non-Benzodiazepine hypnotic drugs within 3 months prior to study initiation.
3. History of Epilepsy and or anti-epileptic drugs.
4. Pregnancy or breast feeding.
5. Clinically relevant ECG abnormalities.
6. History of alcohol or drug abuse within 3 years prior to the screening visit.
7. Known hypersensitivity to drugs of the same class as the study treatment, or any excipients of the drug formulation.
8. Treatment with another investigational drug within 1 month prior to the screening visit.
9. History of severe head injury.
10. Any acute or chronic illness
11. Xerostomia (endogenic or drug induced).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Bioavailability & Bioequivalence study of sublingual CRLS035 (1.1 mg and 2.2 mg) in a single dose administration | 3 months
  To determine the Bioavailability and Bioequivalence of sublingual CRLS035 (1.1 and 2.2 mg) in a single dose administration using the marketed IV flumazenil formulation (0.2 mg) as the comparator [Cmax, Tmax, Cmin, Tmin, AUC0-∞, AUC0-t, T1/2, and F]
Number of participants with adverse events | 3 months
  To determine the number of participants with adverse events to sublingual CRLS035 administration (1.1 mg and 2.2 mg)

SECONDARY OUTCOMES:
Dose Escalation | 3 months
  The secondary objectives are to characterize the concentration time course of two dose levels of SL CRLS035 to support dose selection for Phase 2 and 3 studies and to evaluate number of participants with adverse events and tolerability of flumazenil formulations.
High Fat Diet and Water Consumption effect | 3 months
  To evaluate the effect of high fat diet and water consumption on the PK profile.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel